CLINICAL TRIAL: NCT06609564
Title: Effects of Inspiratory Muscle Training on Respiratory Muscle Strength, Diaphragm Thickness, and Diaphragm Excursion in Mechanically Ventilated Intensive Care Patients
Brief Title: Inspiratory Muscle Training in Mechanically Ventilated Patients in Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Harun Taşkın, Assistant Professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 60116787-020/55139
Record Dates: First submitted 2024-09-16; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Intensive Care Patients Invasively Ventilated; Mechanical Ventilation; Inspiratory Muscle Training; Diaphragm Ultrasonography
Keywords: Physiotherapy and Rehabilitation; Inspiratory Muscle Training; Ultrasound of Diaphragm; Intensive Care Unit; Mechanical Ventilation

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inspiratory Muscle Training (Experimental): Inspiratory muscle training in addition to convantional chest physiotherapy
  Interventions: Device: inspiratory muscle training
- Convational Chest Physiotherapy (Experimental): Diaphragm breathing, costal expansion exercises, postural drainage, effective coughing, in-bed range of motion exercises, and mobilization
  Interventions: Other: Convantional chest physiotherapy

INTERVENTIONS:
Device: inspiratory muscle training — Inspiratory muscle training with a pressure-adjustable device
  Arms: Inspiratory Muscle Training
Other: Convantional chest physiotherapy — Chest physiotherapy
  Arms: Convational Chest Physiotherapy

SUMMARY:
In addition to conventional chest physiotherapy, inspiratory muscle training will be applied in mechanically ventilated intensive care patients. It is aimed to examine the effects of inspiratory muscle training on respiratory muscle strength, diaphragm thickness, and diaphragm excursion in intubated or tracheostomized patients with mechanical ventilation in the intensive care unit.

DETAILED DESCRIPTION:
Subjects who mechanically ventilated in the intensive care unit will be divided two groups. Study group will recieve inspiratory muscle training in addition to convantional chest physiotherapy. Control group will recieve convantional chest physiotherapy. Training will continue until discharge or until the 21st day of the training. Respiratory muscle strength, diaphragm thickness and diaphragm excursion were measured before training and before discharge.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* hemodynamic stability and alert
* able to spontaneously trigger the ventilator and perform at least one command for activation of respiratory muscles
* required mechanical ventilation support with continuous spontaneous ventilation mode or pressure- or volume-controlled intermittent mandatory ventilation (6 breaths/min) mode
* required pressure support ≤ 15 cmH2O and PEEP ≤ 10 cmH2O
* unable to breathe without support for 72 consecutive hours following the resolution of factors leading to respiratory failure
* FiO2 of 0.5 or less
* PaO2 greater than 60 mmHg and capable of sufficient gas exchange

Exclusion Criteria:

* cooperation disorder
* trauma or deformity related to the thorax that affect respiration
* progressive neuromuscular disease
* excessive bronchial secretion (requiring more than one suctioning per hour)
* need for continued sedative or analgesic agents
* use of home-type mechanical ventilation before admission to the hospital
* cardiac, pulmonary, or other conditions leading to impaired stability
* impaired cooperation, compliance, and motivation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strengh | 20 minutes
  Respiratory muscle strength was measured as maximal inspiratory pressure.
Diaphragm thickness | 15 minutes
  Diaphragm thickness was evaluated using ultrasound imaging in two-dimensional B mode (4-13 MHz) performed from the midaxillary level from the right intercostal space with patients sitting in a position as upright as possible. The thickness of the diaphragm was ensured with the superficial probe at end-inspiration (Tins) and end-expiration (Texp).
Diaphragm excursion | 20
  Diaphragm excursion was evaluated at the midaxillary level from the right subcostal area with M-mode (2-5 MHz) ultrasonography in normal inspiration and deep inspiration.

SECONDARY OUTCOMES:
Physical Function in Intensive Care Test (PFIT) | 20 minutes
  The PFIT is a test battery applied by the researchers that consists of four main headings: "Support (from sitting to standing up)," "Cadence (steps/minute)," "Shoulder (flexion strength)," and "Knee (extension strength)." Stand up from sitting was scored according to the degree of help received (0 = without help, 1 = with the help of one person, 2 = with the help of two people). We recorded standstill as the number of steps and the time elapsed while the standing still action was performed. Shoulder and knee muscle strength were assessed using a manual muscle test (0 = no contraction, 1 = contraction only, 2 = movement completed when gravity is eliminated, 3 = movement completed against gravity, 4 = movement completed with less than maximum resistance to gravity, 5 = movement completed with maximum resistance to gravity)
Duration of intubation | 3-15 days
  After the subjects were included in the study duration of intubation was recorded.
Extubation rate | 3-15 days
  Weaning rates of patients from mechanical ventilation
Rate of discharge from the intensive care unit | 8-21 days
  Discharge rate of patients included in the study from intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No